CLINICAL TRIAL: NCT00387374
Title: A Phase II Study of Prophylactic Radiation Therapy for the Prevention of Hemoptysis in Advanced Non Small Cell Lung Cancer in Combination With Bevacizumab, Paclitaxel, and Carboplatin in Patients at High Risk for Bevacizumab-Associated Hemoptysis
Brief Title: Radiation Therapy, Bevacizumab, Paclitaxel, and Carboplatin in Treating Patients With Unresectable Stage IIIB or Stage IV Non-Small Cell Lung Cancer at High Risk for Hemoptysis Caused by Bevacizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02704; CCC-PHII-78; N01CM62208 (NIH); N01CM62201 (NIH); N01CM62203 (NIH); N01CM62209 (NIH); CDR0000504067 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Adenosquamous Cell Lung Cancer; Drug/Agent Toxicity by Tissue/Organ; Hemoptysis; Squamous Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Hemoptysis; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Paclitaxel; Taxes; Carboplatin; Radiotherapy; Radiation

ARMS (2):
- Stratum I (radiotherapy, bevacizumab, chemotherapy) (Experimental): Patients undergo prophylactic radiotherapy on days 1-5 and 8-12. Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes on day 15. Patients also receive paclitaxel IV over 3 hours or carboplatin IV over 30-60 minutes and bevacizumab IV over 30-90 minutes on day 36 (course 2).
  Interventions: Biological: bevacizumab; Drug: paclitaxel; Drug: carboplatin; Radiation: radiation therapy
- Stratum II (radiotherapy, chemotherapy, bevacizumab) (Experimental): Patients undergo prophylactic radiotherapy and receive paclitaxel and carboplatin as in stratum I. Patients also receive bevacizumab IV over 30-90 minutes on day 15 (course 1). In both strata, treatment with paclitaxel, carboplatin, and bevacizumab repeats every 21 days for 5-6 courses in the absence of disease progression or unacceptable toxicity. Patients with complete or partial response or stable disease may continue to receive single-agent bevacizumab every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: paclitaxel; Drug: carboplatin; Radiation: radiation therapy

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation

SUMMARY:
This phase II trial is studying the side effects and how well giving radiation therapy together with bevacizumab, paclitaxel, and carboplatin works in treating patients with unresectable stage IIIB or stage IV non-small cell lung cancer at high risk for hemoptysis caused by bevacizumab. Radiation therapy uses high-energy x-rays to kill tumor cells. It may also prevent hemoptysis caused by bevacizumab. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of non-small cell lung cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with bevacizumab and chemotherapy may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety of prophylactic chest radiotherapy, bevacizumab, paclitaxel, and carboplatin in patients with unresectable stage IIIB or IV non-small cell lung cancer at high risk for bevacizumab-associated hemoptysis.

SECONDARY OBJECTIVES:

I. Assess progression-free survival of patients treated with this regimen. II. Assess the rate of objective response, overall survival, time to response, and response duration in irradiated lesions and non-irradiated lesions in these patients.

OUTLINE: This is an open-label, pilot, multicenter study. Patients are assigned sequentially to 1 of 2 treatment strata.

Stratum I: Patients undergo prophylactic radiotherapy on days 1-5 and 8-12. Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes on day 15. Patients also receive paclitaxel IV over 3 hours or carboplatin IV over 30-60 minutes and bevacizumab IV over 30-90 minutes on day 36 (course 2).

Stratum II: Patients undergo prophylactic radiotherapy and receive paclitaxel and carboplatin as in stratum I. Patients also receive bevacizumab IV over 30-90 minutes on day 15 (course 1). In both strata, treatment with paclitaxel, carboplatin, and bevacizumab repeats every 21 days for 5-6 courses in the absence of disease progression or unacceptable toxicity. Patients with complete or partial response or stable disease may continue to receive single-agent bevacizumab every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 12 months.

PROJECTED ACCRUAL: A total of 72 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed primary non-small cell lung cancer (NSCLC)* meeting the following criteria:

  * Squamous cell or mixed squamous-nonsquamous histology with predominant squamous component (≥ 50% squamous) with a primary, unresected endobronchial lesion

    * No small cell component
  * Centrally located primary tumor, defined by the following:

    * Primary tumor of any T stage within or touching the zone of the proximal bronchial tree

      * Zone is defined as a 3-dimensional volume with a perimeter of 2 cm in each direction around the proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus, right and left lower lobe bronchi)
      * Any disease within this volume must not invade blood vessels determined by a contrast-enhanced CT scan evaluation of the entire thorax with thin slices (≤ 5 mm) through the area of central tumor bulk (i.e., no evidence of vessel invasion radiological evaluation)
* Stage IIIB (with malignant pleural effusion) or stage IV disease

  * Patients with stage IIIB NSCLC without an effusion are eligible if they are not candidates for combined modality therapy with curative intent (i.e., radical chemoradiotherapy)
* At high risk for bevacizumab-associated hemoptysis

  * Hemoptysis estimated as between 2.5 mL and 10 mL (largest volume of single episode of hemoptysis) in the past 2 months
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* No known brain metastases by contrast-enhanced CT scan or gadolinium-enhanced MRI of the brain
* No clinical or radiologic evidence of an existing or impending spinal cord compression
* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Life expectancy > 6 months
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine normal OR creatinine clearance ≥ 50 mL/min
* INR < 1.5
* aPTT ≤ 1.5 times ULN
* No serious medical conditions, including any of the following:

  * Unstable angina
  * Myocardial infarction or stroke (cerebrovascular accident or transient ischemic attack) within the past 6 months
  * Congestive heart failure
  * Active cardiomyopathy
  * Unstable ventricular arrhythmia
  * Symptomatic peripheral vascular disease
  * Active peptic ulcer disease
  * Uncontrolled psychotic disorders
  * Serious infections
  * Other medical conditions potentially aggravated by treatment
* No social situation that would preclude study compliance
* No other active malignancy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* No history of bleeding diathesis or coagulopathy associated with elevated risk of bleeding
* No uncontrolled hypertension (i.e., resting blood pressure consistently higher than systolic > 150 mm Hg and/or diastolic > 100 mm Hg with or without antihypertensive medication), history of labile hypertension, or history of poor compliance with antihypertensive medication
* No clinically significant proteinuria (24-hour urine protein < 1,000 mg)
* No serious or nonhealing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No significant traumatic injury within the past 28 days
* No history of known allergy or reaction attributed to compounds of similar chemical or biological composition to bevacizumab, such as Chinese hamster ovary cell proteins or other recombinant human or humanized antibodies, Cremophor EL®, or other agents used in study treatment
* No pre-existing peripheral neuropathy > grade 1
* No prior thoracic radiotherapy
* At least 12 months since prior chemotherapy

  * No prior chemotherapy for advanced disease
* No prior therapy with angiogenesis, vascular endothelial growth factor (VEGF), or VEGF-receptor inhibitors

  * Cyclooxygenase-2 inhibitors as a noncancer therapy allowed
* At least 28 days since prior and no concurrent major surgery or open biopsy
* At least 12 months since prior anticancer therapy for any other malignancy except basal cell carcinoma of the skin, localized prostate cancer, or in situ carcinoma of the cervix
* At least 10 days since prior therapeutic anticoagulants or therapeutic thrombolytic agents
* No concurrent aspirin (> 325 mg/day) or antiplatelet agents, including dipyridamole, ticlopidine, clopidogrel bisulfate, or cilostazol

  * Other concurrent nonsteroidal anti-inflammatory drugs allowed
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents or therapies

  * Steroids for pain, anorexia, or quality of life allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Safety of treatment as measured by the incidence of grade 3-5 hemoptysis, as assessed by NCI CTCAE version 3.0 | Up to 12 months after completion of treatment
  All toxicities will be tabulated.

SECONDARY OUTCOMES:
Response rate according to RECIST | Up to 12 months
  Estimated with a 95% confidence interval half-width of about 16%. If both stratum are pooled, the response rate will be estimated within 12%.
Overall survival | Up to 12 months
  Calculated based on the method of Kaplan-Meier, and will be presented for each stratum and for the combined results.
Progression-free survival defined as the duration of time from start of protocol treatment to time of progression or death according to RECIST | Up to 2 years
  Calculated based on the method of Kaplan-Meier, and will be presented for each stratum and for the combined results.

CONTACTS AND LOCATIONS:
Overall Officials: Zelanna Goldberg, Principal Investigator — California Cancer Consortium
Locations (1):
- California Cancer Consortium